CLINICAL TRIAL: NCT02165605
Title: Randomized, Double-Blind, Vehicle-Controlled Pilot Study of the Efficacy and Safety of HylaCareTM in the Treatment of Acute Skin Changes in Patients Undergoing External Beam Radiotherapy for Tumors of the Breast.
Brief Title: HylaCare in the Treatment of Acute Skin Changes in Patients Undergoing Radiotherapy for Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Asal Rahimi, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STU 092012-058
Record Dates: First submitted 2013-12-19; First posted 2014-06-17 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: external beam radiotherapy; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HylaCare (Experimental): HylaCare cream Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line. The product and placebo will also be applied to the contra-lateral breast in the same fashion, as a further control. The study drug and placebo will be applied three (3) times daily, but not within 4 hours prior to radiation treatment.
  Interventions: Drug: HylaCare
- Placebo (Placebo Comparator): The patient is her own control.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HylaCare — cream
  Arms: HylaCare
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This will be a randomized, double blind, vehicle-controlled evaluation of the effectiveness and safety of HylaCareTM. The study will employ the patient as her own control, a commonly used method for the evaluation of topical dermatologic agents. Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line. The product and placebo will also be applied to the contra-lateral breast in the same fashion, as a further control. The study drug and placebo will be applied three (3) times daily.

DETAILED DESCRIPTION:
Patients will be allocated to the treatment using a randomized permuted block. There will be no stratification. Patients will be randomized to receive the investigational product to be applied to either the medial (inside) or lateral (outside) portion of the breast, a placebo product will be used on the other side. Patients and clinical investigators will be blinded to the treatment assignments.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 or older
* Diagnosis of breast cancer
* Intact breast (not surgically absent)
* Planned fractionated external beam radiotherapy to be delivered by opposing, tangential beams to 50.4 Gy in 28 fractions with a planned photon or electron boost of 10Gy in 5 fractions (for a total of 33 fractions)
* Ability to understand and comply with the requirements of this study
* Ability to give Informed Consent
* For sexually active females, patient agrees to use acceptable method of birth control

Exclusion Criteria:

* Women who are pregnant or lactating
* Use of concomitant skin care preparations at any of the treated or control portal areas to be observed
* Any infection or unhealed wound of the radiotherapy portal areas, or generalized dermatitis
* Severe renal failure creatinine > 3.0 within 6 months of study registration
* Allergic history, including anaphylaxis or severe allergies to products in study serum or placebo
* Planned relocation which would make follow-up visits impossible during the course of the study
* Collagen vascular disease such as Lupus, or scleroderma

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Rahimi A, Mohamad O, Albuquerque K, Kim DWN, Chen D, Thomas K, Wooldridge R, Rivers A, Leitch M, Rao R, Haley B, Ahn C, Garwood D, Spangler A. Novel hyaluronan formulation for preventing acute skin reactions in breast during radiotherapy: a randomized clinical trial. Support Care Cancer. 2020 Mar;28(3):1481-1489. doi: 10.1007/s00520-019-04957-0. Epub 2019 Jul 4. PMID 31273506

RESULTS

PARTICIPANT FLOW:
Groups:
- HA Serum Vs. Control Cream (Placebo): Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line. The product and placebo will also be applied to the other breast in the same fashion, as a further control. The study drug and placebo will be applied three times daily, but not within 4 hours prior to radiation treatment.
Period: Overall Study
Arm/Group | HA Serum Vs. Control Cream (Placebo)
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hylacare-Experimental: HylaCare cream-Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line. The product and placebo will also be applied to the contra-lateral breast in the same fashion, as a further control. The study drug and placebo will be applied three (3) times daily, but not within 4 hours prior to radiation treatment. The patient is her own control.
Arm/Group | Hylacare-Experimental
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 60 [33 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Acute Skin Toxicity Per NCI-CTC v4.0
Description: NCI-CTC (National Cancer Institute-Common Terminology Criteria) version 4.0 was used to assessed acute skin toxicity grade by physician. Toxicity grade range from Grade 0 to Grade 5, with higher grade indicating worst skin toxicity.
Time Frame: Week 5 during radiation therapy
Population: All 28 patients were assigned to both arms HA formulation (Hylacare study cream) on the medial or lateral half of the irradiated breast and the control cream (placebo) on the other half. Each patient will use both HA study cream and placebo cream on breast receiving radiation treatment.
Measure: Count of Participants; unit: Participants
Groups:
- HylaCare; Placebo: Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line. The product and placebo will also be applied to the contra-lateral breast in the same fashion, as a further control. The study drug and placebo will be applied three times daily, but not within four hours prior to radiation treatment. Each patient will use both HA study cream and placebo.
Arm/Group | HylaCare | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Grade 0 | 3 | 3
  Grade 1 | 19 | 18
  Grade 2 | 6 | 7
  Grade ≥3 | 0 | 0

2. Primary Outcome: Acute Skin Toxicity Per NCI-CTC v4.0
Description: NCI-CTC(National Cancer Institute-Common Terminology Criteria) version 4.0 was used to assessed acute skin toxicity grade by physician. Toxicity grade range from Grade 0 to Grade 5, with higher grade indicating worst skin toxicity.
Time Frame: Week 2 post-radiation therapy
Population: We only analyze available data
Measure: Count of Participants; unit: Participants
Arm/Group | HylaCare | Placebo
Number analyzed (Participants) | 27 | 27
Participants
  Grade 0 | 5 | 3
  Grade 1 | 19 | 23
  Grade 2 | 3 | 1
  Grade ≥ 3 | 0 | 0

3. Primary Outcome: Acute Skin Toxicity Per Investigator Grading Scale
Description: Investigator Grading Scale is used to assessed acute skin toxicity. Score range from grade 0 to 6 with 0 = normal skin
  1. = light epidermal irritation, consisting of the onset of erythema, possibly associated with slight edema
  2. = erythema with dry desquamation
  3. = wet desquamation </= 2 cm
  4. = wet desquamation from 2.1 - 5cm
  5. = wet desquamation from 5.1 - 9 cm
  6. = wet desquamation > 9.1 cm
Time Frame: Week 5 during radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | HylaCare | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Grade 0 | 3 | 4
  Grade 1 | 18 | 14
  Grade 2 | 7 | 10
  Grade ≥ 3 | 0 | 0

4. Primary Outcome: Acute Skin Toxicity Per Investigator Grading Scale
Description: as for outcome 3
Time Frame: Week 2 post-radiation therapy
Population: We only analyzed data that were available
Measure: Count of Participants; unit: Participants
Arm/Group | HylaCare | Placebo
Number analyzed (Participants) | 27 | 27
Participants
  Grade 0 | 4 | 2
  Grade 1 | 13 | 12
  Grade 2 | 10 | 13
  Grade ≥3 | 0 | 0

5. Secondary Outcome: Acute Skin Toxicity, as Measured by Number of Participants With Skin Reactions
Description: Acute skin toxicity, as measured by number of participants with skin reactions via self assessment
Time Frame: Week 5 during radiation therapy
Measure: Count of Participants; unit: Participants
Arm/Group | HylaCare | Placebo
Number analyzed (Participants) | 28 | 28
Participants
  Skin reaction | 13 | 7
  No Skin reaction | 15 | 21

ADVERSE EVENTS:
Time Frame: The independent panel (two radiation oncologists and two breast surgeons) evaluated photographs of the breasts taken at week 5 during and 2 weeks post-RT
Description: Expected adverse event due to radiation with and without the skin cream (Hylacare).
  * Erythema
  * Pain
  * Tenderness
  * Irritability
  * Burning
  * Dryness
  * Hypersensitivity
  * Hair loss
Groups:
- Expected Adverse Events With and Without Skin Cream(Hylacare): Expected adverse event due to radiation with and without the skin cream (Hylacare).
  * Erythema
  * Pain
  * Tenderness
  * Irritability
  * Burning
Arm/Group | Expected Adverse Events With and Without Skin Cream(Hylacare)
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 14/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expected Adverse Events With and Without Skin Cream(Hylacare) (N=28)
Desquamation (Skin and subcutaneous tissue disorders) | 14 (14) — HA serum: 6 participants (21%) Placebo: 8 participants (29%)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2014-05-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT02165605/Prot_000.pdf